CLINICAL TRIAL: NCT00978016
Title: A Dose-Response Efficacy and Safety Study of Arbaclofen Placarbil (XP19986) as Adjunctive Therapy in Subjects With Gastroesophageal Reflux Disease (GERD) Who Are Incomplete Responders to a Proton Pump Inhibitor (PPI)
Brief Title: A Study to Evaluate the Efficacy and Safety of Arbaclofen Placarbil (XP19986) as Adjunctive Therapy in Subjects With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP-B-078
Record Dates: First submitted 2009-09-11; First posted 2009-09-16 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — arbaclofen placarbil; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- arbaclofen placarbil-Cohort 1 (Experimental): arbaclofen placarbil 20 mg QD with PPI*
  * Allowable PPIs : Rabeprazole Sodium 20 mg QD, Esomeprazole Magnesium 20 mg or 40 mg QD, Lansoprazole 15 mg or 30 mg QD, Pantoprazole 20 mg or 40 mg QD, Omeprazole 20 mg or 40 mg QD, Omeprazole/sodium bicarbonate 20 mg or 40 mg QD, Dexlansoprazole 30 mg or 60 mg QD
  Interventions: Drug: arbaclofen placarbil-Cohort 1; Drug: PPI
- arbaclofen placarbil-Cohort 2 (Experimental): arbaclofen placarbil 40 mg QD with PPI*
  * Allowable PPIs : Rabeprazole Sodium 20 mg QD, Esomeprazole Magnesium 20 mg or 40 mg QD, Lansoprazole 15 mg or 30 mg QD, Pantoprazole 20 mg or 40 mg QD, Omeprazole 20 mg or 40 mg QD, Omeprazole/sodium bicarbonate 20 mg or 40 mg QD, Dexlansoprazole 30 mg or 60 mg QD
  Interventions: Drug: arbaclofen placarbil-Cohort 2; Drug: PPI
- arbaclofen placarbil-Cohort 3 (Experimental): arbaclofen placarbil 20 mg BID with PPI*
  * Allowable PPIs : Rabeprazole Sodium 20 mg QD, Esomeprazole Magnesium 20 mg or 40 mg QD, Lansoprazole 15 mg or 30 mg QD, Pantoprazole 20 mg or 40 mg QD, Omeprazole 20 mg or 40 mg QD, Omeprazole/sodium bicarbonate 20 mg or 40 mg QD, Dexlansoprazole 30 mg or 60 mg QD
  Interventions: Drug: arbaclofen placarbil-Cohort 3; Drug: PPI
- arbaclofen placarbil-Cohort 4 (Experimental): arbaclofen placarbil 30 mg BID with PPI*
  * Allowable PPIs : Rabeprazole Sodium 20 mg QD, Esomeprazole Magnesium 20 mg or 40 mg QD, Lansoprazole 15 mg or 30 mg QD, Pantoprazole 20 mg or 40 mg QD, Omeprazole 20 mg or 40 mg QD, Omeprazole/sodium bicarbonate 20 mg or 40 mg QD, Dexlansoprazole 30 mg or 60 mg QD
  Interventions: Drug: arbaclofen placarbil-Cohort 4; Drug: PPI
- Placebo-Cohort 5 (Placebo Comparator): Placebo dose with PPI*
  * Allowable PPIs : Rabeprazole Sodium 20 mg QD, Esomeprazole Magnesium 20 mg or 40 mg QD, Lansoprazole 15 mg or 30 mg QD, Pantoprazole 20 mg or 40 mg QD, Omeprazole 20 mg or 40 mg QD, Omeprazole/sodium bicarbonate 20 mg or 40 mg QD, Dexlansoprazole 30 mg or 60 mg QD
  Interventions: Drug: Placebo-Cohort 5; Drug: PPI

INTERVENTIONS:
Drug: arbaclofen placarbil-Cohort 1 — After the 4 week screening period, eligible subjects will be randomized to adjunctive study treatment (arbaclofen placarbil 20 mg QD) for 7 weeks including titration and taper periods
  Other Names: XP19986
  Arms: arbaclofen placarbil-Cohort 1
Drug: Placebo-Cohort 5 — After the 4 week screening period, eligible subjects will be randomized to adjunctive study treatment (placebo) for 7 weeks including titration and taper periods
  Other Names: XP19986 matching placebo
  Arms: Placebo-Cohort 5
Drug: arbaclofen placarbil-Cohort 2 — After the 4 week screening period, eligible subjects will be randomized to adjunctive study treatment (arbaclofen placarbil 40 mg QD) with for 7 weeks including titration and taper periods
  Other Names: XP19986
  Arms: arbaclofen placarbil-Cohort 2
Drug: arbaclofen placarbil-Cohort 3 — After the 4 week screening period, eligible subjects will be randomized to adjunctive study treatment (arbaclofen placarbil 20 mg BID) for 7 weeks including titration and taper periods
  Other Names: XP19986
  Arms: arbaclofen placarbil-Cohort 3
Drug: arbaclofen placarbil-Cohort 4 — After the 4 week screening period, eligible subjects will be randomized to adjunctive study treatment (arbaclofen placarbil 30 mg BID) for 7 weeks including titration and taper periods
  Other Names: XP19986
  Arms: arbaclofen placarbil-Cohort 4
Drug: PPI — Allowable PPIs : Rabeprazole Sodium 20 mg QD, Esomeprazole Magnesium 20 mg or 40 mg QD, Lansoprazole 15 mg or 30 mg QD, Pantoprazole 20 mg or 40 mg QD, Omeprazole 20 mg or 40 mg QD, Omeprazole/sodium bicarbonate 20 mg or 40 mg QD, Dexlansoprazole 30 mg or 60 mg QD
  Other Names: Proton Pump Inhibitor

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of arbaclofen placarbil (XP19986) versus placebo as adjunctive therapy in subjects with troublesome GERD symptoms despite therapy with approved doses of a Proton Pump Inhibitor (PPI).

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of GERD by a gastroenterologist
2. minimum of 3 months of GERD symptoms prior to screening.
3. currently taking an FDA approved dose of PPI therapy for symptomatic GERD for at least 4 weeks prior to screening
4. experienced partial relief of GERD symptoms while receiving approved dose and regimen of PPI therapy
5. experienced GERD symptoms, defined as heartburn (with or without regurgitation or other GERD symptoms) on ≥ 3 days during the week prior to screening

Exclusion Criteria:

1. evidence of erosive esophagitis or erosive gastritis on upper gastrointestinal endoscopy during screening
2. has not experienced any GERD symptom improvement after an adequate course of PPI treatment (at least 2 weeks)
3. unstable or severe medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Heartburn Episodes | 6 weeks
  number of episodes

SECONDARY OUTCOMES:
Regurgitation Episodes | 6 weeks
  number of episodes

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — XenoPort, Inc.
Locations (61):
- United States (59):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Sherwood, Arkansas
  - Anaheim, California
  - Lancaster, California
  - Mission Hills, California
  - Sacramento, California
  - San Diego, California
  - Stanford, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Lafayette, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Milford, Connecticut
  - Waterbury, Connecticut
  - Jupiter, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Clive, Iowa
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Monroe, Louisiana
  - Shreveport, Louisiana
  - Annapolis, Maryland
  - Hagerstown, Maryland
  - Brockton, Massachusetts
  - Ann Arbor, Michigan
  - Egg Harbor, New Jersey
  - Binghamton, New York
  - Brooklyn, New York
  - Great Neck, New York
  - Johnson City, New York
  - Lake Success, New York
  - Charlotte, North Carolina
  - Fayetteville, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Fargo, North Dakota
  - Columbus, Ohio
  - Norman, Oklahoma
  - Pittsburgh, Pennsylvania
  - Uniontown, Pennsylvania
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Bellaire, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Logan, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Christiansburg, Virginia
  - Waukesha, Wisconsin
- Canada (2):
  - Guelph, Ontario
  - Toronto, Ontario

REFERENCES:
- [Derived] Vakil NB, Huff FJ, Cundy KC. Randomised clinical trial: arbaclofen placarbil in gastro-oesophageal reflux disease--insights into study design for transient lower sphincter relaxation inhibitors. Aliment Pharmacol Ther. 2013 Jul;38(2):107-17. doi: 10.1111/apt.12363. Epub 2013 May 30. PMID 23721547